CLINICAL TRIAL: NCT03710694
Title: A European Multicenter, Randomized, Parallel-group Study to Evaluate the Safety and Efficacy/Performance of DAV132 in Hospitalized Patients at High Risk for Clostridium Difficile Infection and Who Receive Fluoroquinolones for the Treatment of Acute Infections
Brief Title: Safety and Efficacy of DAV132 in Patients at High-Risk for Clostridium Difficile Infection (CDI)
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Da Volterra (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAV132-CL-2001; CIV-18-03-023465 (Other: EUDAMED)
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAV132 group (Experimental): Patients randomized to the DAV132 arm will be administered DAV132 concomitantly with fluoroquinolones.
  Interventions: Device: DAV132
- No DAV132 group (No Intervention): Patients randomized to the No DAV132 arm will receive only fluoroquinolones, according to local standard of care.

INTERVENTIONS:
Device: DAV132 — DAV132:
  * Dosage: 15 g/day activated charcoal (22.5 g/day DAV132)
  * Route: Oral
  * Duration: duration of fluoroquinolone treatment + 2 days
  DAV132 is regulated as a medical device in Europe and as a drug in the United States of America.
  Arms: DAV132 group

SUMMARY:
The purpose of this study is to determine the safe use and evaluate the efficacy/performance of DAV132 in hospitalized patients at high risk for Clostridium difficile infection (CDI) and who receive fluoroquinolones (FQs) for the treatment of acute infections or for prophylaxis of febrile neutropenia.

DETAILED DESCRIPTION:
Da Volterra develops DAV132, a novel therapeutic option preserving the intestinal microbiota, to prevent potentially life-threatening conditions such as CDI or emergence of antibiotic-resistant bacteria. Prevention of CDI remains critical unmet need, especially for patients at high risk of developing such infection.

ELIGIBILITY:
Inclusion Criteria. Eligible patients for the study must meet ALL the following inclusion criteria:

1. Male or female ≥18 years of age
2. Hospitalized patients requiring a systemic antibiotic treatment for a proven or strongly suspected bacterial infection (lower respiratory tract infection [LRTI], complicated urinary tract infection [cUTI]) or prophylactic treatment of febrile neutropenia for neutropenic patient
3. Patients who are intended to receive one of the following FQs: moxifloxacin, levofloxacin, or ciprofloxacin, by oral or parenteral route, for an intended duration of 5 days (minimum) to 21 days (maximum), in monotherapy
4. Patients expected to stay in hospital for at least 3 days after randomization
5. Patients with the following conditions:

   - Previous history of CDI (no more than 2 episodes) within six months prior to study inclusion

   OR

   - Patient aged ≥65 years, and presenting with at least two of the following:
   * Previous cumulated exposure of at least 5 days to any antibiotics within the last 90 days
   * Patients who have at least one concurrent severe comorbidity among the following: malignant disease, chronic renal failure, cardiopulmonary condition (such as chronic congestive heart failure or severe arterial hypertension), diabetes mellitus, or liver cirrhosis
   * Previous hospitalization of more than 72h within the last 90 days, or patient receiving long-term nursing care for more than one month within the last 90 days
6. Female patients participating in the study must be:

   - of non-childbearing potential: surgically sterilized at least 3 months prior to inclusion, or postmenopausal (menopause is defined as being aged >60 years, or aged between 45 and 60 years and being amenorrheic for ≥2 years)

   OR

   - of childbearing potential, and:

   • using an efficient double contraception from inclusion up to 24 hours after the end of the treatment period: hormonal contraception (including patch, contraceptive ring, etc.), intra-uterine device, or other mechanical contraception method

   AND

   condom, or diaphragm or cervical/vault cap, or spermicide

   AND

   must have a negative urine pregnancy test prior to inclusion to the study.
7. Patients who have given their written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria: Eligible patients for this study will be excluded if any of the following conditions are present:

1. Antibacterial treatment within seven days before randomization
2. Fluoroquinolone indication other than LRTI, cUTI, or febrile neutropenia prophylaxis
3. Patients with suspected or diagnosed CDI at screening, and/or receiving a treatment effective against CDI
4. Patients with diarrhea corresponding to Bristol stool chart types 5-7, combined with a stool frequency of at least three stools in 24 or fewer consecutive hours, regardless of its etiology
5. Patients using probiotics for prevention of CDI and refusing to stop them at inclusion and during the study
6. Patients currently taking activated charcoal
7. Patients who have received a fecal microbial transplantation within the last 90 days prior to study screening
8. A critically ill patient for whom transfer to an intensive care unit is scheduled, or patient who may likely have critical clinical deterioration within 48 hours;
9. Patients with serious, uncontrolled disease, including but not limited to neutropenia expected to last >7 days (Investigator discretion) or with an estimated life expectancy shorter than 6 months
10. Patients diagnosed with any cancer requiring taxane-based chemotherapy
11. Patients with digestive stoma, known conditions at risk for intestinal obstruction, or known achlorhydria
12. Contra-indication to oral therapy (eg, severe nausea/vomiting or ileus) or patient having tube feeding
13. Patients unable or expected to be unable within 48 hours to receive a medication by oral route administration
14. Known hypersensitivity to the activated charcoal, or to any of the constituents or excipients of DAV132
15. Patients taking any drug/medication acting on (eg, metronidazole; sulfasalazine) or absorbed in the colon.
16. Female patients planning a pregnancy, pregnant or breastfeeding
17. Patients already included into this study
18. Patients in an exclusion period of a previous study
19. Patients with any social or logistical condition which in the opinion of the Investigator, may interfere with the conduct of the study, such as incapacity to understand well, not willing to collaborate, or cannot easily be contacted after discharge
20. Patients not covered by a health insurance system where applicable and in compliance with the recommendations of the national laws in force relating to biomedical research.
21. Patients under administrative or legal supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Safety endpoint: Proportion of patients having at least one adverse event (AE) related to DAV132 and/or to fluoroquinolones (FQs) and which relationship to product (DAV132 or FQ) is confirmed by the Independent Adjudication Committee (IAC). | 51 days after randomization
  The IAC will review AEs according to the IAC charter, including Clostridium difficile infection (CDI) and antibiotic-associated diarrhea (AAD), in a blinded manner across both treatment groups, and confirm whether each AE is related or not to DAV132 and/or to the FQ received by the patient.

SECONDARY OUTCOMES:
Safety endpoint: Number of AEs and proportion of patients with at least one AE | 51 days after randomization
Efficacy/performance endpoint, clinical:Proportion of patients with CDI | 51 days after randomization
Efficacy/performance endpoint, clinical: Proportion of patients with AAD | 51 days after randomization
Efficacy/performance endpoint, clinical: Plasma levels of FQs | Day 4
Efficacy/performance endpoint, biological: Level of free fecal concentrations of FQs | Day 1, Day 4, Day 6, 10 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Level of α-diversity of the intestinal microbiota | Day 1, Day 6, 10 days after the end of FQs, and 30 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Change from D1 of α-diversity of the intestinal microbiota | Day 6, 10 days after the end of FQs, and 30 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Levels of β-diversity of the intestinal microbiota | Day 6, 10 days after the end of FQs, and 30 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Proportion of patients with resistant bacteria and/or yeasts in feces | Baseline and up to 10 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Proportion of patients with at least one occurrence of resistant bacteria and yeasts in feces (among patients negative at baseline) | up to 10 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator
Efficacy/performance endpoint, biological: Proportion of patients with acquisition of intestinal colonization by C. difficile (among patients negative at baseline) | up to 10 days after the end of FQs
  Duration of treatment with FQs ranges from 5 to 21 days, at the discretion of the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Maria J.G.T Vehreschild, MD, Principal Investigator — Universitaetsklinikum Frankfurt
Locations (29):
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment Sveti Ivan Rilski - Kozloduy EOOD Internal Department, Kozloduy
  - MHAT "Dr Nikola Vasilev " AD 1, Kyustendil
  - MHAT "Dr. Stamen Iliev" AD 4, Montana
  - Pernik EOOD Specialized Hospital for Active Treatment of Pulmonary Diseases - Phthisiatry Department, Pernik
  - Hosp Ruse EOOD, Rousse
  - Multiprofile Hospital for Active Treatment Silistra AD Department of pneumology and phtisiatry, Silistra
  - Military Medical Academy, Clinic of Infectious Diseases, Sofia
  - UMHATEM N.I.Pirogov Department of internal diseases Clinic of internal diseases, Sofia
  - MHAT Sv. Anna Clinic of Urology, Varna
- Germany (4):
  - Universitätskliniken Köln (AöR) Klinik I für Innere Medizin, Cologne
  - Universitaetsklinikum Frankfurt, Medizinische Klinik II, Frankfurt am Main
  - Universitaetsklinikum Jena Klinik für Innere Medizin IV, Jena
  - Medizinische Universitaetsklinik Abteilung Innere Medizin I, Tübingen
- Romania (11):
  - Institutului Clinic Fundeni, Secţia Clinica Urologie III, Bucharest
  - Spitalul Clinic de Boli Infecţioase şi Tropicale Dr. Victor Babeş, Secţia Pneumologie II, Bucharest
  - Spitalului de Boli Infectioase si Tropicale "Dr. Victor Babes" Sectia Clinica de Boli Infectioase si Tropicale VI - adult, Bucharest
  - Institutul de Pneumoftiziologie "MariusNasta" (Pavilionul IV), Sectia Pneumologie VII, Bucharest
  - The Oncology Institute "Prof. Dr. Ion Chiricuţă", Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Secţia Clinică Pneumologie I, Cluj-Napoca
  - Spitalul Clinic de Boli Infecţioase si Pneumoftiziologie Victor Babeş Craiova, Secţia Boli Infecţioase Adulţi II, Craiova
  - Spitalului Universitar de Urgenta Elias, Clinica Universitara de Geriatrie, Gerontologie si Psihogeriatrie, Sos. Bucuresti-Ploiesti, Otopeni
  - Spitalul Clinic de Boli Infecţioase si Pneumoftiziologie "Dr. Victor Babeş" Timişoara, Clinica II Pneumologie, Timișoara
  - Spitalului Clinic de Boli Infecţioase şi Pneumoftiziologie "Dr. Victor Babeş", Secţia Pneumologie II, Timișoara
  - Spitalului Clinic Judeţean de Urgenţă "Pius Brînzeu" Timişoara, Secţia Clinică Urologie, Timișoara
- Serbia (5):
  - Clinical Hospital Centre Bezanijska Kosa Pulmonology Department, Belgrade
  - General Hospital Department for Lung Diseases and Tuberculosis, Čačak
  - Clinical Centre Kragujevac Clinic for Infectious Diseases, Kragujevac
  - Clinical Centre of Nis Clinic for Lung Diseases, Niš
  - Health Centre Uzice Department for Lung Diseases and Tuberculosis, Užice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Gunzburg J, Ducher A, Modess C, Wegner D, Oswald S, Dressman J, Augustin V, Feger C, Andremont A, Weitschies W, Siegmund W. Targeted adsorption of molecules in the colon with the novel adsorbent-based medicinal product, DAV132: A proof of concept study in healthy subjects. J Clin Pharmacol. 2015 Jan;55(1):10-6. doi: 10.1002/jcph.359. Epub 2014 Jul 16. PMID 25042595
- [Background] de Gunzburg J, Ghozlane A, Ducher A, Le Chatelier E, Duval X, Ruppe E, Armand-Lefevre L, Sablier-Gallis F, Burdet C, Alavoine L, Chachaty E, Augustin V, Varastet M, Levenez F, Kennedy S, Pons N, Mentre F, Andremont A. Protection of the Human Gut Microbiome From Antibiotics. J Infect Dis. 2018 Jan 30;217(4):628-636. doi: 10.1093/infdis/jix604. PMID 29186529
- [Background] Burdet C, Sayah-Jeanne S, Nguyen TT, Hugon P, Sablier-Gallis F, Saint-Lu N, Corbel T, Ferreira S, Pulse M, Weiss W, Andremont A, Mentre F, de Gunzburg J. Antibiotic-Induced Dysbiosis Predicts Mortality in an Animal Model of Clostridium difficile Infection. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e00925-18. doi: 10.1128/AAC.00925-18. Print 2018 Oct. PMID 30061286
- [Background] Burdet C, Sayah-Jeanne S, Nguyen TT, Miossec C, Saint-Lu N, Pulse M, Weiss W, Andremont A, Mentre F, de Gunzburg J. Protection of Hamsters from Mortality by Reducing Fecal Moxifloxacin Concentration with DAV131A in a Model of Moxifloxacin-Induced Clostridium difficile Colitis. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00543-17. doi: 10.1128/AAC.00543-17. Print 2017 Oct. PMID 28739791